CLINICAL TRIAL: NCT03193697
Title: Efficacy and Safety of Cemented and Cementless Prostheses in the Repair of Unstable Intertrochanteric Fractures in the Elderly: a Prospective, Single-center, Non-randomized, Controlled, Clinical Trial With 6-month Follow-up
Brief Title: Efficacy and Safety of Cemented and Cementless Prostheses for Unstable Intertrochanteric Fractures in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harrison International Peace Hospital (Other)
Responsible Party: Principal Investigator, Tiemiao Yu, Principal Investigator, Harrison International Peace Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HarrisonIPH_01
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Intertrochanteric Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): Old patients with unstable intertrochanteric fractures underwent total hip arthroplasty. Forty-four patients in the control group received a cemented SPII prosthesis (Link, Germany).
  Interventions: Device: cemented SPII prosthesis
- trial group (Experimental): Old patients with unstable intertrochanteric fractures underwent total hip arthroplasty. Forty-two patients in the trial group received cementless Wagner prosthesis (Zimmer, USA).
  Interventions: Device: cementless Wagner prosthesis

INTERVENTIONS:
Device: cemented SPII prosthesis — Old patients with unstable intertrochanteric fractures underwent total hip arthroplasty. Forty-four patients in the control group received a cemented SPII prosthesis (Link, Germany).
  Other Names: control group
  Arms: control group
Device: cementless Wagner prosthesis — Old patients with unstable intertrochanteric fractures underwent total hip arthroplasty. Forty-two patients in the trial group received cementless Wagner prosthesis (Zimmer, USA).
  Other Names: trial group
  Arms: trial group

SUMMARY:
This trial explores the application of different hip replacement materials in elderly patients with unstable intertrochanteric fracture, and aims to provide the experience and basis for hip arthroplasty in elderly osteoporosis patients with unstable intertrochanteric fracture.

DETAILED DESCRIPTION:
Background Intertrochanteric fractures are common types of hip fractures. With the growth of the global aging population, the elderly fracture patients with osteoporosis are increasing. Thus, the difficulty of treating intertrochanteric fractures increases accordingly. Unstable intertrochanteric fractures refer to the fractures from femoral neck base to lesser trochanter level. With the continuous development of China's aging trend, the number of aging population is increasing gradually; the incidence of unstable intertrochanteric fractures is increasing year by year. Clinically, more than 90% of intertrochanteric fractures occur in the elderly over 65 years of age, and the mortality rate is at a high level. Patients with unstable intertrochanteric fractures are older, and body function gradually degrades. The reduction and fixation of this disease are difficult. Therefore, early to find timely and effective treatment is of great significance to patients with unstable intertrochanteric fractures.

Clinically, internal fixation and artificial joint replacement are the primary methods of treating unstable intertrochanteric fractures. The surgical approach of internal fixation is easily affected by the bone quality of the patients. If the patient has different degrees of osteoporosis, it will lead to the failure of the first operation, affecting the prognosis of the patient. Therefore, this kind of operation method is not accepted gradually in clinical practice. The efficacy of joint replacement for treatment of intertrochanteric fracture is remarkable. It can make the patient obtain the immediate stability and reduce complications, so it is very popular with the patients and physicians in the clinic. The most commonly used artificial joint replacement materials in clinic have two types: cemented and cementless prostheses, but the difference in their efficacies and safeties remains poorly understood.

Adverse events To record adverse events, including incision pain, bone cement poisoning, pulmonary infection, mental disorders and acute cerebral infarction.

If severe adverse events occurred, investigators reported details, including the date of occurrence and measures taken to treat the adverse events, to the principle investigator and the institutional review board within 24 hours.

Data collection, management, analysis and open-access Data collection: Records of all cases reported in the trial were complete, clear and true. The case reports were consistent with the patient's original data and the declared data. The collected data were input to the computer in the record room of Harrison International Peace Hospital.

Data management: Data were processed by a special person, and aggregated once a month. During clinical trials, hospital clinic visits were conducted periodically by the clinical ombudsman to ensure that all the contents of the protocols were strictly observed. Simultaneously, raw data were checked to ensure the consistency with the case report form.

Data analysis: Statistical analysis was performed by professional statisticians. The statisticians wrote the research report and submitted it to the researcher for review.

Data open-access: Anonymized trial data will be published at www.figshare.com.

Statistical analysis Statistical analysis was performed using SPSS 19.0 software (IBM, Armonk, NY, USA) and followed the intention-to-treat principle.

Normally distributed measurement data were expressed as means ± standard deviation and minimums and maximums. Non-normally distributed measurement data were expressed as the lower quartile (q1) and median and upper quartiles (q3). Count data were expressed as the percentage. Two-sample t-test was performed for comparison of Harris hip scores, operation time, intraoperative blood loss, postoperative blood transfusion volume, ambulation time and postoperative amount of drainage in both groups. Repeated measures analysis of variance was conducted for intragroup comparison of Harris hip scores at various time points. Pearson X2 test was carried out for comparison of excellent and good rate of Harris hip scores and incidence of adverse reaction in both groups.

The significance level was α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Unstable intertrochanteric fractures identified by imaging and laboratory examination
* Age: Greater than 65 years old
* Irrespective of sex
* Volunteered to participate in this test, and signed informed consent

Exclusion Criteria:

* Replacement contraindications, such as acute myocardial infarction
* Obvious obstacles in language communication and communication

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Harris hip scores | at postoperative 6 months
  To assess the recovery of hip function.The number of patients with excellent and good Harris hip scores/total number of patients × 100%. High excellent and good rate indicates good hip function.

SECONDARY OUTCOMES:
X-ray | Changes from preoperative 6 months to postoperative 6 months
  To observe morphological changes in the hip.Morphology of the hip was observed in the anteroposterior and lateral images. Heterotopic ossification was classified via the Brooker classification system.

IPD SHARING:
Plan to Share IPD: Undecided